CLINICAL TRIAL: NCT00509860
Title: A Phase II Study of Irinotecan (Camptosar) in Patients With Advanced Sarcomas
Brief Title: Irinotecan (Camptosar) in Patients With Advanced Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM03-0002
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Sarcoma
Keywords: Advanced Sarcomas; Irinotecan; Camptosar; CPT-11
MeSH Terms: conditions — Sarcoma | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irinotecan (Experimental): Irinotecan 16 mg/m2 by vein daily over 1 hour for 5 Days
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — 16 mg/m2 by vein Daily Over 1 Hour x 5 Days
  Other Names: Camptosar; CPT-11

SUMMARY:
Primary Objectives:

1. To determine the efficacy of the topoisomerase I (topo I) inhibitor irinotecan, delivered via a low-dose protracted schedule to patients with advanced sarcoma.
2. To determine the toxicity profile of irinotecan, using a protracted schedule, in this pretreated patient population.

DETAILED DESCRIPTION:
Irinotecan is a chemotherapy drug that fights cancer by interfering with the cancer cells' ability to divide and grow.

Before treatment starts, you will be asked questions about your health and have a complete physical exam. You will have an electrocardiogram (ECG - a test that measures the electrical activity of the heart). You will have computed tomography (CT) scans and x-rays to check on the status of the disease. If your doctor feels it is necessary, you may also have a magnetic resonance imaging (MRI). Women who are able to have children must have a negative blood or urine pregnancy test.

During treatment, you will receive irinotecan by vein over one hour, once a day for 5 days in a row. This will be followed by 2 days of no study drug treatment, then 5 more days of treatment with irinotecan. This 12-day period will be followed by 9 days of rest (no study drug). This 21-day period is called a cycle of therapy. You will continue to receive treatment (cycles repeated) as long as the disease does not get worse or until maximal shrinkage of the cancer. Treatment may be taken on an outpatient basis.

During treatment, you will have blood collected (1-2 teaspoons) once a week for routine tests. At least once every cycle of treatment (3 weeks) you will have a physical exam and be asked questions about you health.

After the first 2 cycles, the disease will be re-evaluated. You will have blood tests (1-2 teaspoons), x-rays, and CT scans. If your doctor feels it is necessary, you may also have a MRI. This re-evaluation will be repeated every 4 cycles.

If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

Your doctor may choose to follow up with long-term exams at his/her discretion.

This is an investigational study. Irinotecan is FDA approved and is commercially available. Up to 60 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of all ages.
2. Patients must have histologic proof of a sarcoma.
3. Patients must have locally advanced / metastatic disease that is inoperable or incurable with surgery.
4. If patient has a history of prior malignancy, there must be histologic documentation that metastatic disease is sarcoma.
5. Patients must have received or refused standard chemotherapy for disease.
6. Patients must have at least one lesion that is clearly defined, measurable or objectively evaluable. This lesion cannot have been previously irradiated unless progression has been demonstrated after radiation.
7. Patients must have a life expectancy of at least 12 weeks and a Zubrod performance status of < 2.
8. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of this hospital. The only approved consent form is appended to this protocol.
9. Patients must receive no other concurrent chemotherapy or immunotherapies. Patients must have recovered from any previous chemotherapy. They must have been off treatment at least 4 weeks from the previous chemotherapy (6 weeks for stem cell toxins) and have recovered from any side effects or toxicity prior to the institution of irinotecan.
10. Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte counts of at least 1000/cubic mm and platelet count of at least 50,000/cubic mm determined within 2 weeks prior to the first treatment.
11. Patients should have adequate hepatic function with a bilirubin < 2 times the upper limit of normal, and Serum glutamic pyruvic transaminase (SGPT) < 3 times the upper limit of normal determined within 2 weeks prior to the first treatment.

Exclusion Criteria:

1. Pregnant or lactating women will be excluded, due to unknown side effects on the fetus.
2. Patients with severe pulmonary insufficiency will be excluded.
3. Patients of childbearing potential not willing to utilize birth control during and for at least 3 months following completion of the trial shall not be eligible.
4. Patients with an overt psychosis or mental disability, those with psychological or social situation that would interfere with study follow-up, or otherwise incompetent to give informed consent shall be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-03; Primary Completion 2007-08 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of the topoisomerase I (topo I) inhibitor irinotecan, delivered via a low-dose protracted schedule to patients with advanced sarcoma | Four 3-week cycles (12 weeks)
  Efficacy based on dose limiting toxicity (DLT). Unacceptable toxicity is defined as grade 3 or 4 nonhematologic toxicity, or if expressed by the patient as unacceptable despite the grade. Patients evaluated for toxicity at the end of each cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Benjamin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org